CLINICAL TRIAL: NCT00479648
Title: A Phase II, Double-Blind, Randomised, Controlled, Multi-Centre Study to Evaluate the Immunogenicity, Safety and Tolerability of Three Formulations of CSL412 in Adults (≥ 18 to ≤ 45 Years) and Older Adults (≥ 60 Years)
Brief Title: A Phase 2 Study of Immunogenicity, Safety and Tolerability of CSL412 in Elderly Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CSLCT-IIV-06-27
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Active Comparator): Inactivated trivalent influenza vaccine
  Interventions: Biological: Inactivated trivalent influenza vaccine
- 2 (Experimental): CSL412 formulation
  Interventions: Biological: CSL412
- 3 (Experimental): CSL412 formulation
  Interventions: Biological: CSL412
- 4 (Experimental): CSL412 formulation
  Interventions: Biological: CSL412

INTERVENTIONS:
Biological: CSL412
  Arms: 2; 3; 4
Biological: Inactivated trivalent influenza vaccine
  Arms: 1

SUMMARY:
Current influenza vaccines have a reduced efficacy in the elderly. This study will investigate the immunogenicity, safety and tolerability of an adjuvanted influenza vaccine in elderly participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 to ≤ 45 OR ≥ 60
* Ability to provide pre-vaccination venous blood sample

Exclusion Criteria:

* History of clinically significant medical conditions
* Immunomodulative therapy
* Acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
seroprotection rate, HI titre & seroconversion/ significant increase
grade 3 or higher, vaccine associated fever or vaccine associated site ulceration, abscess or necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hancox, Dr, Principal Investigator — Chiltern International
Locations (1):
- Chiltern International, Slough, United Kingdom